CLINICAL TRIAL: NCT02319226
Title: Toward Immune Biomarkers for Tolerance and GvHD in Humans
Acronym: BioGvHD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Other Study IDs: PRTSN1339002N
Record Dates: First submitted 2014-12-13; First posted 2014-12-18 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Bone Marrow Transplantation; Graft vs Host Disease; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Transplantation from an HLA-identical sibling donor — The study will include a cohort of 60 patients transplanted from an HLA-identical sibling donor.

SUMMARY:
Graft-versus-Host Disease (GVHD), is the most frequent and severe complication of allogeneic hematopoietic stem cell transplantation (HSCT). Much of our knowledge on the pathophysiology of GVHD has been gained from experimental models but far less from the study of the disease in humans. Recent developments in basic biology open new avenues to the development of biomarker sets that could predict GVHD severity and prognosis that could be tested and validated through well-designed multicenter clinical trials.

The main goal of this project is to further our understanding of the pathogenic mechanisms of human GVHD on one hand, and of functional immune tolerance on the other. Furthermore, this study aims at setting up a clinically relevant biomarker set in human GVHD and immune tolerance in a discovery cohort.

The objectives of this project are:

1. To define phenotypic, functional and molecular correlates of acute GVHD early after HSCT/at its onset 2. To study thymic reconstitution and the T-cell repertoire after HSCT during period 2 3. To identify functional and molecular correlates of immune tolerance in long-term survivors of HSCT 4. Preparing for biomarker validation into a clinical trial We propose a prospective analysis of a cohort of 680 patients transplanted from an HLA-identical sibling donor at Saint Louis hospital. Analyses will be performed during 3 critical, clinically relevant, periods.

1. Period 1: Analysis at the onset of GVHD, or at the time of engraftment 30 days after HSCT in patients not developing GVHD. An additional blood sample will also be analyzed 90 days after HSCT.
2. Period 2: Thymic function analysis using measurements of T-cell receptor excision circles (TREC) will be performed at 6 and 12 months post-transplant for all patients. T-cell receptor analysis on sorted T-cell populations will be performed by NGS.
3. Period 3: In "tolerant" patients (patients more than 2 years after HSCT not requiring immunosuppressive treatment), or in patients still requiring immunosuppressive therapy after 2 years. We will also analyze the corresponding immune parameters for each donor.

The longitudinal design of this study will allow us to provide an integrated view of GVHD pathophysiology and mechanisms of immune tolerance in human.

Prospectively identified phenotypic, molecular or functional biomarkers will then be tested, in a subsequent study, from biological materials prospectively collected within the French wide CryoStem cohort. Thus, as the final task of this project, we will perform statistical analyses taking into account confounding clinical variables influencing the outcome (i.e. GVHD-related death or tolerance). Preparing for a clinical trial will need moving from classical Bioinformatics analyses into clinically relevant statistical analyses that include sequential biological measurement in the discovery set cohort. Main points that will be taken into accounts for this task are the followings;

1. Transplant-related mortality (TRM) can be estimated in the range of 20%; 2year post-allogeneic HSCT
2. TRM is mostly (even if totally) due to GVHD and its associated immune deficiency
3. GVHD cumulative incidence can be estimated in the range of 40%
4. 80 patients will be prospectively studied and 30 patients will be analyzed (cross sectional study) for part 3 only.
5. Since GVHD-related mortality and tolerance are mutually exclusive situation the optimal calculation for the validation cohort can be expected
6. This calculation will be the basis for the proposal of an interventional clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients transplanted from an HLA-identical sibling donor

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients transplanted from an HLA-identical sibling donor
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2019-02 (Actual); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
acute Graft-versus-Host Disease (GVHD) early after allogeneic hematopoietic stem cell transplantation (HSCT) | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital siant-Louis, Paris, France